CLINICAL TRIAL: NCT02231463
Title: Influence of Two Different PEEP Niveaus and a Trendelenburg Positioning Manoeuvre on Subclavian Vein Diameter as a Surrogate Parameter in Punctures of Central Veins
Brief Title: Influence of Two Different PEEP Niveaus and a Trendelenburg Positioning Manoeuvre on Subclavian Vein Diameter
Status: Withdrawn | Type: Observational
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Principal Investigator, Jochen Hinkelbein, PD Dr. med., Universitätsklinikum Köln
Other Study IDs: CVL-Position-1
Record Dates: First submitted 2014-06-04; First posted 2014-09-04 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Insufficiency; Cardiac, Complicating Surgery
Keywords: ultrasound
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ultrasound measurement: measuring subclavian vein Diameter in six Groups:
  neutral positioning, PEEP 0 cm H2O, neutral positioning, PEEP 5cm H2O, neutral positioning, PEEP 10cm H2O, Trendelenburg positioning -20°, PEEP 0 cmH2O, Trendelenburg positioning -20°, PEEP 5 cmH2O, Trendelenburg positioning -20°, PEEP 10 cmH2O After these measurements a central venous catheter is used to measure the central venous pressure.
  Interventions: Other: neutral positioning, PEEP 0 cm H2O; Other: neutral positioning, PEEP 5cm H2O; Other: neutral positioning, PEEP 10cm H2O; Other: Trendelenburg positioning -20°, PEEP 0 cmH2O; Other: Trendelenburg positioning -20°, PEEP 5 cmH2O; Other: Trendelenburg positioning -20°, PEEP 10 cmH2O

INTERVENTIONS:
Other: neutral positioning, PEEP 0 cm H2O — neutral positioning, PEEP 0 cm H2O
Other: neutral positioning, PEEP 5cm H2O — neutral positioning, PEEP 5cm H2O
Other: neutral positioning, PEEP 10cm H2O — neutral positioning, PEEP 10cm H2O
Other: Trendelenburg positioning -20°, PEEP 0 cmH2O — Trendelenburg positioning -20°, PEEP 0 cmH2O
Other: Trendelenburg positioning -20°, PEEP 5 cmH2O — Trendelenburg positioning -20°, PEEP 5 cmH2O
Other: Trendelenburg positioning -20°, PEEP 10 cmH2O — Trendelenburg positioning -20°, PEEP 10 cmH2O

SUMMARY:
In 50 Patients who are undergoing a planned surgical procedure which require a central venous catheter the diameter of the subclavian vein is measured by ultrasound under 6 different conditions.

DETAILED DESCRIPTION:
In 50 Patients who are undergoing a planned surgical procedure which require a central venous catheter the diameter of the subclavian vein is measured by ultrasound under 6 different conditions. The conditions are

1. neutral positioning, PEEP 0 cm H2O,
2. neutral positioning, PEEP 5cm H2O,
3. neutral positioning, PEEP 10cm H2O,
4. Trendelenburg positioning -20°, PEEP 0 cmH2O,
5. Trendelenburg positioning -20°, PEEP 5 cmH2O,
6. Trendelenburg positioning -20°, PEEP 10 cmH2O After these measurements a central venous catheter is used to measure the central venous pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* cardiosurgery or neurosurgery
* written informed consent
* ECG: inus rhythm

Exclusion Criteria:

* peacemaker
* kontraindications for PEEP
* pulmonary disease
* hemodynamically instable patients
* pregnancy
* pulmonal Hypertension
* ejection fraction < 35%
* severe valvular disease
* tricuspid insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a operative procedure which requires a central venous catheter
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Diameter of vein | only 1 day (the day of the measurement); no follow-up is required
  measurement of vein Diameter by ultrasound in a randomized order

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Hinkelbein, MD, Principal Investigator — UK Köln
Locations (1):
- UK Köln, Cologne, North Rhine-Westphalia, Germany